CLINICAL TRIAL: NCT00210977
Title: An Observational Study of Subjects Treated With Erythropoietin Receptor Agonists for Anemia Who Developed Anti-erythropoietin Antibodies
Brief Title: A Study of Patients Treated With Erythropoietin Receptor Agonists for Anemia Who Developed Anti-erythropoietin Antibodies
Status: Withdrawn | Type: Observational
Why Stopped: The study never started due to zero enrolment
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR003277; EPO-IMU-302 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Anemia
Keywords: Anemia; Erythropoietin; Epoetin alfa; Erythropoietin receptor agonist (ERA) therapy; Anti-erythropoietin antibodies (anti-EPO Ab); Recombinant human erythropoietin; Pure red cell aplasia; Darbepoetin
MeSH Terms: conditions — Anemia; Arthritis, Juvenile; Red-Cell Aplasia, Pure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for pharmacogenomic analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Erythropoietin receptor agonist: Participants with borderline serum anti erythropoietin (EPO) antibody (Ab) titers and who are treated with any erythropoietin receptor agonist (ERA) for any indication, having anti-EPO Ab identified by radioimmunoprecipitation (RIP), who are responding to ERA therapy, will be included in the study.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. All participants will be maintained on their regular dose regimen of standard-of-care treatment, under the guidance of the treating physician/investigator.

SUMMARY:
The purpose of this study is to assess the presence of anti erythropoietin antibodies (anti EPO Ab) in participants responding to any erythropoietin receptor agonist (ERA) therapy to treat or prevent anemia without loss of effectiveness to see if they will develop pure red cell aplasia or loss of effectiveness to recombinant erythropoietin and to measure the duration of effectiveness of ERA therapy.

DETAILED DESCRIPTION:
This is an observational (study in which the investigators/physicians observe the participant's data and measure their outcomes), international, multicenter (study conducted at multiple sites), cohort (group of individuals with similar characteristics) study. The study consists of prestudy phase, observational phase (2 years), and follow-up phase (1 year). Approximately 50 participants who already receiving ERA therapy for anemia will be observed in this study. In the observational phase, participants' erythropoietin antibody status (positive or negative), clinical progress, treatment for anemia or prevention of anemia, and outcome will be monitored. During this study, enrolled participants will continue to receive standard-of-care treatment for their disease from their individual investigators as before enrollment to this study. Safety evaluations will include assessment of adverse events which will be monitored throughout the study. The total duration of the study will be 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Receiving any ERA therapy for any cause of anemia and having responded to the ERA therapy for at least 3 months
* Positive or borderline serum for antibodies to erythropoietin identified by serum radioimmunoprecipitation
* Maintained a stable hemoglobin within a 3-month period that has not decreased more than 2 g/dL in any 1-month period and with no increase in red blood cell transfusion requirement
* An ERA maintenance dose that has not increased more than 50 percentages from initial effective dose
* If blood count information is available, must have a count of reticulocytes (immature red blood cells) greater than or equal to 30 million/L

Exclusion Criteria:

* Stem cell or bone marrow transplantation
* Treatment with medication that decreases the ability of the immune system to function normally, within the last 3 months
* Participants who have shown a loss of effectiveness to ERA therapy, defined as participants who initially responded to treatment for anemia [a rise in hemoglobin which lasted for a minimum of 3 months] followed by an unexplained decrease in hemoglobin (greater than or equal to 2 g/dL) within a 1-month period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with positive or borderline serum anti erythropoietin antibody titer and who are responding to any erythropoietin receptor agonist (ERA) therapy for any cause of anemia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-12; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Presence of Anti-Erythropoietin Antibodies (anti-EPO Ab) | Up to 2 years
  An antibody is a large Y-shaped protein secreted into the blood and is used by the immune system to identify and neutralize foreign objects such as bacteria and viruses. Presence of anti-EPO Ab will help to find out participant's progress to the outcomes loss of effectiveness, suspected pure red cell aplasia, or confirmed pure red cell aplasia.
Duration of Effectiveness of Erythropoietin Receptor Agonist Therapy | Up to 2 years

SECONDARY OUTCOMES:
Concentration of Plasma Anti Erythropoietin Antibody | Up to 2 years
Factors That Forecast Progression to Loss of Effectiveness | Up to 2 years
Factors That Forecast Progression to Suspected Pure Red Cell Aplasia | Up to 2 years
Factors That Forecast Progression to Confirmed Pure Red Cell Aplasia | Up to 2 years
Number of Participants With Adverse Events | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.